CLINICAL TRIAL: NCT00574366
Title: A Phase I/II Trial of an Oral MTOR Protein Kinase Inhibitor (Everolimus, RAD001) in Combination With an Oral EGFR Tyrosine Kinase Inhibitor (Erlotinib, Tarceva™) In Patients With Metastatic Breast Cancer
Brief Title: Erlotinib and Everolimus in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0523; VU-VICC-BRE-0523; NCT00179270 (obsolete NCT alias)
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Erlotinib Hydrochloride; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib/RAD001 Ph I (Experimental): Tarceva (OSI-774; erlotinib) Everolimus (RAD001)
  Study did not progress to Phase II:
  Experimental: Erlotinib/RAD001 Phase II Maximum tolerated dose of erlotinib (Tarceva,OSI-774) and RAD001 (Everolimus)
  Interventions: Drug: erlotinib; Drug: RAD001

INTERVENTIONS:
Drug: erlotinib — Levels:
  * 1 Erlotinib 50 mg/d
  * 2 Erlotinib 50 mg/d
    * 1 Erlotinib 100 mg/d
    * 2 Erlotinib 100 mg/d
    * 3 Erlotinib 150 mg/d
    * 4 Erlotinib 150 mg/d
  Other Names: Tarceva (OSI-774)
Drug: RAD001 — Levels
  minus 1: RAD001 2.5 mg/d
  minus 2: RAD001 2.5 every other day
  1. RAD001 2.5 mg per day
  2. RAD001 5 mg per day
  3. RAD001 10 mg per day
  4. RAD001 10 mg per day
  Other Names: everolimus

SUMMARY:
RATIONALE: Erlotinib and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erlotinib together with everolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving erlotinib together with everolimus and to see how well it works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of everolimus given in combination with erlotinib hydrochloride in patients with metastatic breast cancer (phase I).
* To determine the antitumor activity of the combination (phase II).
* Determine the rate of clinical benefit (complete response + partial response + stable disease for at least 6 months) in patients with metastatic breast cancer (phase II).

Secondary

* To determine the time to progression.
* To determine PTEN, pAkt, pP70S6K1 and pEGFR in primary tumors at baseline.

OUTLINE: This is an open-label, dose escalation phase I study followed by an open-label phase II study.

* Phase I: Patients receive escalating doses of oral everolimus and oral erlotinib hydrochloride once daily until the maximum tolerated dose (MTD) is determined. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Once the MTD is reached, the recommended dose to be used in the phase II portion of the study is identified.
* Phase II: Patients receive oral everolimus and oral erlotinib hydrochloride as in phase I at the recommended phase II dose determined in phase I.

Patients undergo tissue collection to evaluate tumor levels of PTEN, pAkt, pP70S6K1, and pEGFR at baseline in order to identify predictors of therapeutic response.

After completion of study treatment, patients are followed every 3 months for 2 years (from study entry), every 6 months for 3 years, and annually thereafter.

NOTE: Phase I completed. Investigator did not proceed with Phase II

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast
* Evaluable metastatic disease (no need for measurable disease)
* Must have had anthracycline therapy in the adjuvant setting or failed anthracycline treatment in the metastatic setting

  * Total cumulative dose of lifetime exposure of doxorubicin not greater than 360 mg/m^2 or epirubicin not greater than 640 mg/m^2
* Must have failed previous taxane (paclitaxel or docetaxel) therapy, defined as:

  * Taxane use in the adjuvant setting with metastatic relapse within 12 months of therapy
  * Progression on taxane therapy in the metastatic setting
  * Discontinuation of taxane therapy in the metastatic setting secondary to lack of resolution of ≥ grade 2 toxicity
* No symptomatic brain metastases

  * Patients with a history of brain metastases are eligible provided they are clinically stable and not taking steroids or therapeutic anticonvulsants that are CYP3A4 modifiers
  * Patients with asymptomatic brain metastasis are eligible provided they are not on prophylactic anticonvulsants that are CYP3A4 modifiers
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria

* Menopausal status not specified
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.5 times ULN
* Albumin > 30 g/L
* Creatinine ≤ 1.5 upper limit of normal
* INR normal provided the patient is not on warfarin therapy
* Not pregnant or nursing
* Negative pregnancy test for premenopausal patients
* Fertile patients must use effective barrier method contraception during and for 3 months after completion of study treatment
* Patients must be disease-free of prior invasive cancers for > 5 years with the exception of basal cell or squamous cell cancer of the skin or cervical carcinoma in situ

Exclusion criteria

* Serious or non-healing active wound, ulcer, or bone fracture
* Known human immunodeficiency virus positivity
* Uncontrolled intercurrent illness including, but not limited to, any of the following

  * Ongoing or active infection requiring parenteral antibiotics
  * Impairment of lung function (COPD, lung conditions requiring oxygen therapy)
  * Symptomatic congestive heart failure (New York Heart Association class III or IV heart disease)
  * Unstable angina pectoris or myocardial infarction within the past 6 months
  * Uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg or diastolic blood pressure > 100 mm Hg, found on two consecutive measurements separated by a 1-week period despite adequate medical support)
  * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment)
  * Uncontrolled diabetes
  * Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary

PRIOR CONCURRENT THERAPY:

Inclusion criteria

* See Disease Characteristics
* Prior trastuzumab (Herceptin®) in the first-line treatment of metastatic breast cancer is required for patients who have HER2/neu overexpressing tumors
* More than 6 months since prior cardiac angioplasty or stenting
* Use of endocrine therapy (i.e., aromatase inhibitors, fulvestrant, tamoxifen or ovarian ablation) in the first-line treatment of metastatic breast cancer is required for patients who have estrogen receptor and or progesterone receptor expressing tumors

  * Concurrent endocrine therapy is not allowed
* Patients may receive concurrent radiotherapy to painful bone metastases or areas of impending bone fracture as long as radiotherapy is initiated prior to study entry

  * Patients who have received prior radiotherapy must have recovered from toxicity induced by this treatment
* More than 3 weeks since prior chemotherapy, biological or hormonal therapy while on protocol therapy.
* No other concurrent antineoplastic or antitumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy

Exclusion criteria

* More than 3 prior chemotherapy treatments in the metastatic setting

  * This restriction does not include endocrine therapies or single agent biologic therapies (i.e., trastuzumab [Herceptin®])
* Use of steroids or immunosuppressants
* Use of CYP3A4 modifiers
* Concurrent therapy with trastuzumab (Herceptin®)
* Use of growth support factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], recombinant erythropoietin) during the phase I portion of the study
* Other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-12; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of RAD001 given in combination with erlotinib (Phase I) | at 4 weeks
  MTD will be the dose level at which fewer than 2 of 6 (or 33% of) patients experience dose limiting toxicity (DLT), starting at first 4 weeks.
Anti-tumor activity of RAD001 in combination with erlotinib (Phase II) | at 6 months
  Clinical benefit based upon number of patients with complete response (CR), partial response (PR), and stable disease (SD). Responses are determined by Response Evaluation in Solid Tumors (RECIST)criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions

SECONDARY OUTCOMES:
Time to progression (Phase II) | from study entry to disease progression
  Duration of time to progression of disease.

OTHER OUTCOMES:
To determine PTEN, pAkt, pP70S6K1 and pEGFR in primary tumors at baseline. | at day one
  Breast tissue paraffin-embedded blocks from patients's pre-treatment diagnostic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee